CLINICAL TRIAL: NCT05598372
Title: The Effect of Two Different Methods on Infant Pain During Vaccination and Maternal Anxiety: a Randomized Controlled Study
Brief Title: Infant Pain During Vaccination and Maternal Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-88012460-050.01.04-208074
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-06

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- shotblocker (Experimental): infant pain during vaccination and mother anxiety
  Interventions: Behavioral: shotblocker
- lullaby (Experimental): infant pain during vaccination and mother anxiety
  Interventions: Behavioral: lullaby
- CONTROL (No Intervention): not infant pain during vaccination and mother anxiety

INTERVENTIONS:
Behavioral: shotblocker — infant pain during vaccination and mother anxiety
  Arms: shotblocker
Behavioral: lullaby — infant pain during vaccination and mother anxiety
  Arms: lullaby

SUMMARY:
This research was planned to determine the effect of two different methods on infant pain during vaccination and mother anxiety.The study was planned as a randomized controlled trial. The universe of this research consists of parents and their babies who come to Hocabey Family Health Center in Erzincan Center to receive the hepatitis B dose between these dates according to the vaccination calendar. In this study, it is planned to apply shotblocker and lullaby.

DETAILED DESCRIPTION:
Type of Study The study was planned as a randomized controlled trial. Population and Sample The universe of this research consists of parents and their babies who come to Hocabey Family Health Center in Erzincan Center to receive the hepatitis B dose between these dates according to the vaccination calendar.

Data Collection Tools Demographic Data Form, Neonatal Pain Scale and State Anxiety Scale Newborn Infant Pain Scale (NIPS): The scale used in the assessment of newborn pain consists of 6 categories. It was developed in 1993 and its validity and reliability in our country was made in 1999. The score obtained from the scale varies between 0-7. Scale ; It consists of five behavioral indicators including facial expression, arm movement, leg movement, crying, alertness, and a physiological indicator that includes breathing.

State Anxiety Inventory: The State Anxiety Scale was developed in 1970, and its Turkish validity and reliability study in our country was conducted in 1994. There are a total of 40 statements in the scale. The first twenty items measure the level of anxiety related to the situation, and each statement is "Not at all" (1), "Somewhat" (2), "Very"(3), "Totally"(4). Reverse coded items; Items 1, 2, 5, 8, 10, 11, 15, 16, 19, 20. Points are added and subtracted according to the reverse and direct coded items in the scale. He states that 0-19 points obtained from the scale mean no anxiety, 20-39 points mean mild, 40-59 points mean moderate, 60-79 points mean severe anxiety, and individuals with a score of 60 and above need professional help.

Data Collection Ethics and institutional permissions After the data is received, it will be explained to the participants that the confidentiality of the data will be protected, that personal information will not be requested, that the study is on a voluntary basis, and they will be informed that they can terminate the study at any time. Adolescents who agree to participate in the study will fill in the data collection form, which will take approximately 10 minutes, based on personal notification.

Experimental process In this study, it is planned to apply shotblocker and lullaby. Shotblocker application is not a drug application, it is a small apparatus that performs the blocking process on peripheral nerves to reduce the pain with protruding shape. There is no harm in the application. Another application planned in the study is lullaby. In this application, it is aimed to reduce the baby's pain, which is the painful process, by making the mother who is closest to the baby sing a lullaby. It is very important to compare these two methods. Namely; The effectiveness of two natural and artificial applications will be compared. The fact that this study has not been done before will also provide an important data source to the literature. The planned study will be conducted with 30 lullabies, 30 shotblockers, and 30 babies who come to Hocabey Family Health Center to receive their 6th month Hepatitis B dose and their mothers as a control group to help measure the effectiveness of these two groups. In order to reduce the variables in the application, the nurse who performed the application will be kept constant. For the preliminary application, the principal researcher will be at the center for 1 week and will make observations.

Analysis of the data The data will be evaluated as a result of statistical analyzes using the SPSS package program in computer environment. Descriptive statistics will be displayed as numbers, percentages, and mean±standard deviation. Skewness and Kurtosis values will be checked if the data is suitable for normal distribution. ±1.5 will be taken as the normal distribution limit value. Chi-square test, variance analysis and Pearson correlation analysis will be used in the analysis of the variables. Statistical significance level will be accepted as p˂0.05 in all analyzes.

Research Ethics During the collection of research data, the principle of informed consent, the principle of respect for autonomy and the protection of confidentiality and confidentiality will be followed.

ELIGIBILITY:
Inclusion Criteria:

* The child does not have a disorder in the cognitive developmental area.
* It is time to apply the hepatitis B vaccine of the 6th month.
* Parent giving consent to participate in the study voluntarily and for their child to participate.

Exclusion Criteria:

* The child has a disorder in the cognitive developmental area.
* Failure to apply the 6th month hepatitis B vaccine.
* Parent's voluntarily participating in the study and not giving consent for the child's participation.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Newborn Infant Pain Scale (NIPS) | 9 MONTHS
  The scale used in the assessment of newborn pain consists of 6 categories. It was developed in 1993 and its validity and reliability in our country was made in 1999. The score obtained from the scale varies between 0-7. Scale ; It consists of five behavioral indicators including facial expression, arm movement, leg movement, crying, alertness, and a physiological indicator that includes breathing.
State Anxiety Inventory | 9 MONTHS
  The State Anxiety Scale was developed in 1970, and its Turkish validity and reliability study in our country was conducted in 1994. There are a total of 40 statements in the scale. The first twenty items measure the level of anxiety related to the situation, and each statement is "Not at all" (1), "Somewhat" (2), "Very"(3), "Totally"(4). Reverse coded items; Items 1, 2, 5, 8, 10, 11, 15, 16, 19, 20. Points are added and subtracted according to the reverse and direct coded items in the scale. She states that 0-19 points obtained from the scale mean no anxiety, 20-39 points mean mild, 40-59 points mean moderate, 60-79 points mean severe anxiety, and individuals with a score of 60 and above need professional help.

CONTACTS AND LOCATIONS:
Overall Officials: ARZU SARIALİOĞLU, PHD, Study Director — Ataturk University
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED